CLINICAL TRIAL: NCT01191307
Title: Assess Specific Kinds of Children Challenges for Neurologic Devices Study
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: Carlos Pena, PhD, MS (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Carlos Pena, PhD, MS, Senior Science Policy Advisor, Food and Drug Administration (FDA)
Organization: Food and Drug Administration (FDA) (U.S. Federal Agency)
Other Study IDs: 09-006C
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Primary Dystonia; Epilepsy; Hydrocephalus; Bladder Control; Hearing Impaired (Partially)
Keywords: Primary dystonia; Epilepsy; Hydrocephalus; Bladder Control; Deaf or Hearing Impaired
MeSH Terms: conditions — Dystonic Disorders; Epilepsy; Hydrocephalus; Hearing Loss

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Shunt Implant: hydropcephalus cohort
- Cochlear Implant: hearing impaired cohort
- Spinal Cord Stiumulation: spinal cord injury cohort
- Vagus Nerve Stimulation: epilepsy cohort
- Deep Brain Stimulation: dystonia cohort

SUMMARY:
The ASK CHILDREN study is intended to aid in future development of various neurologic devices (i.e. neuroprostheses). The ASK CHILDREN study seeks to use study information obtained to identify more efficient strategies in the evaluation and review of neuroprostheses regulated by the Agency.

DETAILED DESCRIPTION:
The ASK CHILDREN study is intended to aid in future development of various neurologic devices (i.e. neuroprostheses). The ASK CHILDREN study seeks to use study information obtained to identify more efficient strategies in the evaluation and review of neuroprostheses regulated by the Agency. Specific aims of the clinical study include: (1) Collecting qualitative and quantitative self-report clinical data (through interviews) from children undergoing treatment related to human factors, safety, usability, and adverse events in patients ages 7 to 15 years old implanted with a neuroprosthesis targeting the brain or spinal cord (at two 6 month intervals); and (2) Establish a science-based framework of recommendations based upon the data collected in the ASK CHILDREN Study to help develop more efficient strategies in evaluating pediatric neuroprostheses regulated by the Agency.

ELIGIBILITY:
Primary Dystonia Inclusion Criteria

* Between ages 7 and 15 years of age;
* Implanted Medtronic Activa® Dystonia Therapy (approved or cleared by FDA for pediatric use).
* Neurologic device implanted within the past 12 months;
* Signed assent form document from the child
* Signed permission form from the parent/guardian); and

Exclusion Criteria

* Participation in another clinical investigation that could be jeopardized by participation in the current study;
* Children with severe cognitive impairments (such as children with head injuries resulting in severe cognitive impairment) may be excluded because they may not be capable of self-reporting procedures.
* Unable to comply with terms of the study

Epilepsy Inclusion Criteria

* Between ages 12 and 15 years of age;
* Neurologic device implantation or surgical (in-hospital) adjustment within the past 12 months;
* NeuroCybernetic Prosthesis (NCP®) System (approved or cleared by FDA for pediatric use; the NCP® System is approved for children in ages 12 years and older).
* Signed assent form document from the child; and
* Signed permission form from the parent/guardian).

Epilepsy Exclusion Criteria

* Participation in another clinical investigation that could be jeopardized by participation in the current study; and
* Children with severe cognitive impairments (such as children with head injuries resulting in severe cognitive impairment) may be excluded because they may not be capable of self-reporting procedures.6
* Unable to comply with terms of the study

Pediatric Hydrocephalus Inclusion Criteria

* Between ages 7 and 15 years of age;
* Implanted traditional or adjustable hydrocephalus shunt implant (approved or cleared by FDA for pediatric use).
* Neurologic shunt implantation or surgical (in-hospital) adjustment within the past 12 months;
* Signed assent form document from the child
* Signed permission form from the parent/guardian)

Pediatric Hydrocephalus Exclusion Criteria

* Participation in another clinical investigation that could be jeopardized by participation in the current study; and
* Children with severe cognitive impairments (such as children with head injuries resulting in severe cognitive impairment) may be excluded because they may not be capable of self-reporting procedures.6
* Unable to comply with terms of the study

Spinal Cord Injury Inclusion Criteria

* Between ages 14 and 15 years of age;
* Vocare® Bladder System implant (approved or cleared by FDA for pediatric use).
* Neurologic device implanted within the past 12 months;
* Signed assent form document from the child
* Signed permission form from the parent/guardian); and

Spinal Cord Injury Exclusion Criteria

* Participation in another clinical investigation that could be jeopardized by participation in the current study; and
* Children with severe cognitive impairments (such as children with head injuries resulting in severe cognitive impairment) may be excluded because they may not be capable of self-reporting procedures.
* Unable to comply with terms of the study

Deaf or Hearing Impaired Inclusion Criteria

* Between ages 7 and 15* years of age;
* Implanted cochlear implant (approved or cleared by FDA for pediatric use) with any device adjustment related to device performance or routine care of their current device within the past 12 months;
* Signed assent form document from the child
* Signed permission form from the parent/guardian); and

Deaf or Hearing Impaired Exclusion Criteria

* Participation in another clinical investigation that could be jeopardized by participation in the current study; and
* Children with severe cognitive impairments (such as children with head injuries resulting in severe cognitive impairment) may be excluded because they may not be capable of self-reporting procedures.
* Unable to comply with terms of the study

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary Dystonia Criteria; Between ages 7 and 15 years of age, Approved medical device for Primary Dystonia, Neurologic device implanted within the past 12 months. Epilepsy Criteria; Between ages 12 and 15 years of age; Neurologic device implantation or surgical (in-hospital) adjustment within the past 12 months; Approved medical device. Pediatric Hydrocephalus Criteria; Between ages 7 and 15 years of age, Approved medical device, Neurologic shunt implantation or surgical (in-hospital) adjustment within the past 12 months. Spinal Cord Injury Criteria; Between ages 14 and 15 years of age, Approved medical device, Neurologic device implanted within the past 12 months. Deaf or Hearing Impaired Criteria; Between ages 7 and 15* years of age, Approved medical device.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos L Pena, PhD, Principal Investigator — Food and Drug Administration (FDA)

IPD SHARING:
Plan to Share IPD: No
Data sharing will occur via publication.